CLINICAL TRIAL: NCT04474873
Title: SHOULD THE ERECTOR SPİNAE PLANE BLOCK BE APPLIED IN THE PAIN MANAGEMENT OF PERCUTANOUS NEPHROLITOTOMY SURGERY?
Brief Title: Effectivenes of Erector Spinae Plane Block in Percutaneous Nephrolithotomy?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, semih başkan, assistant professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E1-20-315
Record Dates: First submitted 2020-06-28; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Pain; Nephrolithotomy, Percutaneous; Erector Spinae Plane Block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1:Conventional intravenous analgesia (No Intervention): Conventional intravenous analgesia applied according to surgeon's preference
- Group 2:ESPB (Active Comparator): A 6-13 MHz linear probe was used for ultrasound-guided ESPB (Logiq e, General Electric, USA,) performed at the T11 level. The transverse process was detected by sliding the transducer 3-4 cm laterally from the midline, and after identification of the transverse process, a 20-gauge 100mm insulated echogenic needle (Vygon locoplex, France) was used
  Interventions: Procedure: erector spinae block

INTERVENTIONS:
Procedure: erector spinae block — we administer 15 cc of 0.5% bupivacaine between the erector spine muscle and the transverse process. The distribution of bupivacain was observed on ultrasound.
  Arms: Group 2:ESPB

SUMMARY:
This study investigates the effectiveness of the erector spinae plane block (ESPB) in pain management of patients undergoing PNL.

DETAILED DESCRIPTION:
Although percutaneous nephrolithotomy(PNL) is a minimally invasive procedure, it causes severe postoperative pain due to dilatation of the renal capsule and parenchymal duct and peritubal distension of the nephrostomy tube. PNL-related pain has a limited response to oral and intravenous treatments. The primary aim of our study is to investigate the effectiveness of the erector spinae plane block (ESPB) in pain management of patients undergoing PNL.

Our secondary aim is determining if any possible clinical effect of ESPB in terms of serial peak expiratory flow measurements, postoperative agitation score of the patient (Riker Score), ambulation time, length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing PNL between 18-65 years old

Exclusion Criteria:

* serious cardiac, respiratory, hepatic, renal or haemotologic disease
* mental disorder and hearing problem
* anxiety, depression and / or other psychiatric disorders
* pregnancy
* refusal of patient
* Allergy or contraindications to drugs used in the study
* ASA > 2 Inflammation or infection over injection site Obese patients BMI ≥35/

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | postoperative 24 hours
  the amount of pain that a patient feels ranges across a continuum from none(0) to an extreme amount of pain(10) on a chart.
Dynamic Visual Analog Scale | postoperative 24 hours
  the amount of pain during mobilization, deep breathing or coughing that a patient feels ranges across a continuum from none(0) to an extreme amount of pain(10) on a chart
Peak Expiratory Flow Rate( PEFR) | postoperative 24 hours
  maximum speed of expiration as measured with a peak flow meter

SECONDARY OUTCOMES:
Time for first analgesic requirement | 24 hours
  Time between end of surgery and patients first analgesic demand
ambulation time | 5 days
  first postoperative mobilization time of the patient
length of hospital stay | 1 week
  day of hospitalization
Rikert Agitation Scale | 24 hours
  postoperative agitation score
  1. unarousable
  2. very sedated
  3. sedated
  4. calm and cooperative
  5. agitated
  6. very agitated
  7. dangerous agitation
nausea and vomiting | 24 hours
  incidence of nausea and vomiting
patient satisfaction with anesthesia and analgesia | 24 hour
  4 Likert scale ( the level of satisfaction of a patient ranges from satisfied (1) to nonsatisfied(4)
starting oral intake | 48 hours
  first oral intake
urinary catheter releated pain score(Visual Analog Scale) | postoperative 24 hours
  the amount of pain that a patient feels ranges across a continuum from none(0) to an extreme amount of pain(10) on a chart.
surgeon satisfaction with anesthesia and analgesia | 24 hour
  4 Likert scale ( the level of satisfaction of surgeon ranges from satisfied (1) to nonsatisfied(4)

CONTACTS AND LOCATIONS:
Overall Officials: Semih Baskan, 2, Study Director — Ankara City Hospital Anesthesiology Department
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ibrahim M, Elnabtity AM. Analgesic efficacy of erector spinae plane block in percutaneous nephrolithotomy : A randomized controlled trial. Anaesthesist. 2019 Nov;68(11):755-761. doi: 10.1007/s00101-019-00673-w. Epub 2019 Oct 16. PMID 31620856